CLINICAL TRIAL: NCT06026384
Title: Development and Evaluation of Theory Guided Narrative and Non-narrative Interventions to Enhance Cancer Literacy and Cancer Prevention Beliefs in the Population: a Pilot Study
Brief Title: Evaluation of Text or Animation-based Narrative and Non-narrative Interventions to Enhance Cancer Literacy: a Pilot Study (CLARO)
Acronym: CLARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University of Music, Drama, and Media Hannover (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLARO Pilot; 70114759 (Other Grant/Funding Number: German Cancer Aid)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Cancer Prevention
Keywords: Cancer; Cancer Literacy; Informational Intervention; Health Communication
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-Narrative Text (Experimental): A short text (480 words) that deals with the preventability of cancer cases. It shows that lifestyle factors such as smoking, unhealthy diet, obesity and physical inactivity are responsible for about 40% of cancer cases. It also suggests ways to reduce the risk of cancer through behavioural changes in these areas. A special focus is on nutrition and physical activity. The text was developed on the basis of the Protection Motivation Theory.
  Interventions: Other: text in non-narrative form
- Narrative Text (Experimental): The narrative text contains the same information as the non-narrative text, except that it is built into a story. This makes the text slightly longer at 725 words. The text is about a main character and two work colleagues who share their personal experiences about nutrition and exercise.
  Interventions: Other: text in narrative form
- Non-Narrative Animation (Experimental): The animation with a total duration of 3:12 min is based on the text in non-narrative form and aims to be as fully comparable as possible.
  Interventions: Other: animated video in non-narrative form
- Narrative Animation (Experimental): The animaion (3:45 min) is based on the text in narrative form and aims to be as fully comparable as possible.
  Interventions: Other: animated video in narrative form

INTERVENTIONS:
Other: text in non-narrative form — Participants will be asked to read a text and give feedback afterwards
  Arms: Non-Narrative Text
Other: text in narrative form — Participants will be asked to read a text and give feedback afterwards
  Arms: Narrative Text
Other: animated video in non-narrative form — Participants will be asked to watch a video and give feedback afterwards
  Arms: Non-Narrative Animation
Other: animated video in narrative form — Participants will be asked to watch a video and give feedback afterwards
  Arms: Narrative Animation

SUMMARY:
The goal of this interventional pilot study is to test and evaluate different information materials created to heighten participants cancer literacy, cancer prevention beliefs, and subsequent intention for behavioral changes. Forty individuals, intended to cover a broad socioeconomic background, will participate in the pilot study. Based on the results of this pilot study, the information materials will be adapted for the following main study.

DETAILED DESCRIPTION:
CLARO aims to answer the question, how information materials should be designed to strengthen optimistic beliefs on cancer prevention and to indirectly facilitate the acquisition of cancer literacy.

Four different information materials were developed and will be tested in this pilot study (2x2-design: text or animation-based / narrative or non-narrative). Participants will take part in a 30- to 40-minute survey. As part of the study, they will be randomly assigned to one of the information materials, and asked to evaluate it in depth, both quantitatively and qualitatively. The interviews will be conducted individually and face to face.

Recruitment: Two research assistants will approach potential participants at a shopping center in Heidelberg, Germany, to invite them to participate in the study. Participants will receive a leaflet with further details and contact information. Those interested will be able to participate immediately at a designated room next to the center, provided by the National Cancer Prevention Center, where all interviews will take place, or schedule an appointment via email. As an incentive, participants will receive 30€ via bank transfer upon completing the interview.

Randomization Procedure: Simple randomization - a research assistant will use an Excel spreadsheet to generate random participant codes, which will then be integrated into LimeSurvey to ensure a closed survey environment. The list of codes will be password protected and not accessible to the two research assistants who will conduct the interviews. LimeSurvey will then assign individual codes to participants. Participant codes and allocation details will then be printed on paper and placed within sealed envelopes. Interviewers will then use these envelopes to select the corresponding intervention guide.

Semi-Structured Interview: Post-intervention, participants will take part in a semi-structured interview. With participant permission, all interviews will be audio-recorded on VLC media player. The interviews will be conducted by two research assistants with a background in psychology and previous training on the interview technique.

Transcription: The audio recordings will be transcribed verbatim by the two research assistants using the MAXQDA 2022 (VERBI Software, 2021) and will be reviewed by the principal investigators for accuracy. The interviews, original transcriptions, and data analysis will be in German. All quotes will be translated into English and back-translated by two independent members of the research team to ensure that the meaning will be preserved.

By using a mixed method approach the study will combine quantitative and qualitative methods addressing the following research questions:

Quantitative:

* What is the sample's socio-demographics? (e.g. age, gender, highest educational degree, current occupational status, and income)
* Has there already been personal contact with people with cancer (e.g. through own cancer or cancer in the family)?
* What is the level of engagement in health behaviours (smoking, healthy eating, exercise, BMI)?
* How strongly are Cancer Prevention Beliefs and Cancer Information Overload represented?
* How much do the participants like the material shown? (three questions on satisfaction with the material as well as possible counter-argumentation in order to exclude distortions due to social desirability)
* Can the people in the narrative conditions identify with the characters shown?

Qualitative:

* Do the participants like the materials?
* Is there something wrong with the quality of the materials? (e.g., quality of sound & images, presentation of animated figures, font size, readability...)
* Are the materials comprehensible?
* Is the amount of information appropriate? If not, is it too less or too much?
* Is the information given convincing?
* What are the most important insights gained from the materials? Do any of the information have novelty value?
* Are the given recommendations perceived as helpful?
* Are there ways to improve the materials?
* Might anyone feel excluded or offended by the information?

An inductive content analysis will be carried out to analyse the qualitative data obtained.

The results of the CLARO pilot study will help to improve the intervention materials that will be used for the subsequent main study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years old
* Being able to speak and understand german

Exclusion Criteria:

- Not being able and willing to provide informed consent and complete questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the materials | 20 minutes
  Participants will be asked questions regarding the material presented (qualitatively and quantitatively) covering general satisfaction, comprehensibility, persuasion, affective reactions and potential ways to improve the material.
  The quantitative items regarding general satisfaction and counter-argumentation are rated on a 5-point Likert scale ranging from 1 = "Do not agree at all" to 5 = "Fully agree" with higher scores indicating higher satisfaction with the material as well as higher counter-argumentation.
  Identification with characters will be measured using one item asking "What was the extent to which you could identify with the main characters in the animation?". Participants in the narrative condition will rate this question per character on a scale of 1 (very low) to 10 (very high), so higher scores indicate higher identification.

SECONDARY OUTCOMES:
Cancer Prevention Beliefs & Cancer Information Overload | 5 minutes
  Participans will be assessed asking for agreement with three statements that have been used in previous studies: "It seems like everything causes cancer," "There's not much you can do to lower your chances of getting cancer," and "There are so many recommendations about preventing cancer, it's hard to know which ones to follow". Participants will indicate agreement on a 4-point likert scale ranging from 1 = "strongly agree" to 4 = "strongly disagree".

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center; Alexander Haussmann, Dr., Principal Investigator — German Cancer Research Center; Florian Herbolsheimer, Dr., Principal Investigator — German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No